CLINICAL TRIAL: NCT04695509
Title: The Influence of Propofol Sedation on Neuromediators Concentration
Brief Title: Sedation and Neuromediators Concentration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 502
Record Dates: First submitted 2020-12-18; First posted 2021-01-05 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2020-12

CONDITIONS: Moderate Sedation; Deep Sedation
Keywords: Sedation; Neuromediators

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- moderate sedation (Experimental): patients with American Society of Anesthesiologists (ASA) I-II, Montreal cognitive assessment test ≥ 26, trauma surgery under regional anesthesia with moderate propofol sedation
  Interventions: Drug: moderate propofol sedation (Bispectral index monitoring 70-90; The Richmond Agitation and Sedation scale (RASS) "-2" - "-3"
- deep sedation (Experimental): Arm Description: patients with American Society of Anesthesiologists (ASA I-II), Montreal cognitive assessment test ≥ 26, trauma surgery under regional anesthesia with deep propofol sedation
  Interventions: Drug: deep propofol sedation (BIS 60-70, The Richmond Agitation and Sedation scale (RASS) "-4")

INTERVENTIONS:
Drug: moderate propofol sedation (Bispectral index monitoring 70-90; The Richmond Agitation and Sedation scale (RASS) "-2" - "-3" — Two peripheral venous blood catheters are placed after admission in the operation room and venous blood sample is taken (10 ml). Complete monitoring of vital functions is provided (pulse oximetry, noninvasive blood pressure, electrocardiography, bispectral index monitoring). Doctor anesthesiologist performs regional anesthesia and propofol light-moderate sedation starts. The second blood sample (10 ml) is taken 35-40 minutes after the start of propofol sedation. The third blood sample (10 ml) is taken after emergence from propofol sedation (10-15 minutes after propofol discontinuation). Blood samples are centrifuged and received plasma is frozen at a temperature of -20 C*. After 26 patients are recruited, the blood plasma is analyzed by conducting the enzyme-linked immunosorbent assay (ELISA) of neuromediators (Dopamine, serotonin, Gamma-aminobutyric acid (GABA), acetylcholine, noradrenaline).
  Arms: moderate sedation
Drug: deep propofol sedation (BIS 60-70, The Richmond Agitation and Sedation scale (RASS) "-4") — Two peripheral venous blood catheter is placed after admission in the operation room and venous blood sample is taken (10 ml). Complete monitoring of vital functions is provided (pulse oximetry, blood pressure, electrocardiography, bispectral index monitoring). Doctor anesthesiologist performs regional anesthesia and propofol deep sedation starts. The second blood sample (10 ml) is taken 35-40 minutes after the start of propofol sedation. The third blood sample (10 ml) is taken after emergence from propofol sedation (10-15 minutes after propofol discontinuation). Blood samples are centrifuged and received plasma is frozen at a temperature of -20 C*. After 26 patients are recruited, the blood plasma is analyzed by conducting enzyme-linked immunosorbent assay (ELISA) of neuromediators (Dopamine, serotonin, Gamma-aminobutyric acid (GABA), acetylcholine, noradrenaline).
  Arms: deep sedation

SUMMARY:
Propofol (Propofol Kabi, Registration number from the State Register of Medicines - 000875) is a widely used intravenous anesthetic. It is well known about different effects of propofol infusion, including euphoria, psycholalia, disinhibition, talkativeness, satisfaction etc. However, the basic mechanisms of such effects remain unknown. We suppose that propofol sedation with various levels of sedation (from light to deep) leads to neuromediators changes. We examine dopamine, noradrenaline, acetylcholine, GABA and serotonin in peripheral venous blood before, during and after propofol sedation. Therefore, we suppose drugs for sedation, in particular, propofol will affect neuromediators concentration.

DETAILED DESCRIPTION:
The study is a prospective, nonrandomized, single center investigator design. Twenty-six healthy patients undergoing elective trauma surgery (arthroscopy, reconstructive foot surgery, osteosynthesis of intra-and periarticular fractures of the proxymal humerus) under regional anesthesia (spinal anesthesia or brachial plexus block) with medical propofol sedation are enrolled in this study. Montreal cognitive assessment test is a high validity test for detecting cognitive impairment before operation. American Society of Anesthesiologists (ASA) physical status classification system is used to assess the physical status of patients before operation. Hospital Anxiety and Depression Scale (HADS) is used to determine the levels of anxiety and depression before operation. Two 18 or 20 G venous cannulae are inserted in the left and/or right forearm for drug infusion and blood sampling. The Richmond Agitation and Sedation scale (RASS) and bispectral index monitor A-2000XP (BIS, Aspect Medical Systems, Inc. (USA), Registration certificate for a medical device RZN 2005/498) are used to determine the levels of sedation. Briefly (less than 10 seconds) awakens with eye contact to voice or any movement (but no eye contact) to voice, bispectral index values 70-90 correspond light-moderate sedation. No response to voice, but any movement to physical stimulation, bispectral index monitoring values 60-70 correspond deep sedation. BBraun Space with target control infusion sedation (TCIS, B. Braun Melsungen AG, Registration certificate for a medical device RZN 2013/905) is used for dosing of propofol with moderate (1-st group) or deep sedation (2-nd group). Philips Monitor IntelliVue MP40 (Medizin Systeme Boblingen GmbH, Germany, Registration certificate for a medical device RZN 2014/2009) is used for monitoring the electrocardiogram (ECG), noninvasive blood pressure (NIBP), pulse oximetry during the infusion of the propofol and 15-20 minutes thereafter. Peripheral venous blood samples are taken for analyzing neuromediators concentration 5 minutes before sedation (10 ml), after 35-40 min of propofol sedation (10 ml) and 10-15 minutes after the end of propofol infusion (emergence from sedation). The blood is centrifuged for at least 8 minutes at 4000 revolutions per minute (RPM) in the test tube 367525-BD VACUTAINER (Becton Dickinson), plasma is taken, which is further frozen at a temperature of -20 C in the test tube 363706-BD MICROTAINER (Becton Dickinson). After 26 patients are recruited, the blood plasma is analyzed by conducting the enzyme-linked immunosorbent assay (ELISA, IBL Hamburg) of neuromediators (dopamine (Catalog № Re59161), serotonin (Catalog № Re59121), gamma-aminobutyric acid (GABA), acetylcholine (Catalog № Re59161), noradrenaline (Catalog № Re59261)). Concentrations of neuromediators between moderate and deep sedation groups are compared using Student's t-test for independent samples. Concentrations of neuromediators before, during and after sedation are compared using Friedman-test for dependent samples. All data is presented as mean ± SD, a value of P less than 0.05 is taken as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥ 18 years
* Elective trauma surgery (arthroscopy, reconstructive foot surgery, osteosynthesis of intra-and periarticular fractures of the proxymal humerus) under regional anesthesia (spinal anesthesia or brachial plexus block) with propofol sedation
* Montreal cognitive assessment test ≥ 26
* Patients with American Society of Anesthesiologists (ASA) I-II

Non-inclusion criteria:

* Not written informed consent
* Age˂18 years
* Allergy to sedation drugs
* Pregnancy
* Epilepsy anamnesis
* II-III degree atrioventricular block
* Montreal cognitive assessment test ˂ 26
* Patients with American Society of Anesthesiologists (ASA) ˃ II
* The presence of psychiatric disorders
* Сancer patients with a life expectancy of less than two years

Exclusion Criteria:

* Patient refuse from further participation
* Transition from sedation to general anesthesia
* Allergy on anesthesia drugs during perioperative period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Dopamine concentration changes during moderate and deep sedation | 2 months for each patient from venous blood sampling to enzyme-linked immunosorbent assay (ELISA) dopamine conducting
  Venous blood sampling and enzyme-linked immunosorbent assay (ELISA) are used to evaluate the influence of medical sedation on dopamine concentration
Serotonin concentration changes during moderate and deep sedation | 2 months for each patient from venous blood sampling to enzyme-linked immunosorbent assay (ELISA) serotonin conducting
  Venous blood sampling and enzyme-linked immunosorbent assay (ELISA) are used to evaluate the influence of medical sedation on serotonin concentration
GABA concentration changes during moderate and deep sedation | 2 months for each patient from venous blood sampling to enzyme-linked immunosorbent assay (ELISA) GABA conducting
  Venous blood sampling and enzyme-linked immunosorbent assay (ELISA) are used to evaluate the influence of medical sedation on GABA concentration
Acetylcholine concentration changes during moderate and deep sedation | 2 months for each patient from venous blood sampling to enzyme-linked immunosorbent assay (ELISA) acetylcholine conducting
  Venous blood sampling and enzyme-linked immunosorbent assay (ELISA) are used to evaluate the influence of medical sedation on acetylcholine concentration
Noradrenaline concentration changes during moderate and deep sedation | 2 months for each patient from venous blood sampling to enzyme-linked immunosorbent assay (ELISA) noradrenaline conducting
  Venous blood sampling and enzyme-linked immunosorbent assay (ELISA) are used to evaluate the influence of medical sedation on noradrenaline concentration

SECONDARY OUTCOMES:
Target control infusion (TCI) values of propofol sedation | intraoperative period
  Bbraun Perfusor Space is used for target control propofol infusion. TCI values for moderate sedation are 1,0-2 mcg/ml, deep sedation 2,5-3,5 mcg/ml.
Richmond agitation and sedation scale (RASS) scores | intraoperative period
  RASS is measured during propofol infusion and the target scores for moderate sedation are "-1" - "-3", deep sedation "-4"
Bispectral index monitoring (BIS) values during moderate and deep sedation | intraoperative period
  BIS-monitor А-2000XP (Aspect Medical Systems, USA) is used for evaluating the level of sedation. BIS values for moderate sedation are 70-90, deep sedation 60-70

CONTACTS AND LOCATIONS:
Locations (1):
- City Clinical Hospital № 31 of the Department of Health of Moscow, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available 11/01/2021

REFERENCES:
- See also: Related Info — https://lomonosov-msu.ru/archive/Lomonosov_2020/data/19419/112756_uid128092_report.pdf
- See also: Related Info — https://istina.msu.ru/conferences/presentations/327241590/